CLINICAL TRIAL: NCT00318409
Title: Pilot Study of Acceptability of Bupropion Treatment for Methamphetamine Dependence Among Men Who Have Sex With Men.
Brief Title: Acceptability of Pharmacologic Treatment for Methamphetamine Dependence Among MSM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Public Health Foundation Enterprises, Inc. (Other)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Medical Director, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21DA021090-1; R21DA021090 (NIH)
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Substance Abuse; HIV Infections
Keywords: Methamphetamine; HIV
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Active Comparator): buproprion XL 300mg daily
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): placebo 300mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion
  Other Names: Wellbutrin
  Arms: Bupropion
Drug: Placebo
  Arms: Placebo

SUMMARY:
Studies demonstrate that methamphetamine (meth) use is associated with high-risk sexual behavior among MSM, putting meth-using MSM at extraordinarily high risk for transmitting or acquiring HIV. No studies have tested the feasibility and acceptability of conducting pharmacologic interventions to reduce meth use and meth-associated sexual risk behavior among MSM. The purpose of this pilot study is to determine the feasibility enrolling and retaining meth-dependent MSM into a pharmacologic study of bupropion vs. placebo and measuring the tolerability of and adherence to medication among these participants.

DETAILED DESCRIPTION:
The high rate of meth use among MSM is paralleled by evidence of rises in sexual risk behavior and HIV infection among this population. The MSM meth epidemic, and its link with HIV transmission, underscores the need to pilot test new, innovative modalities to reduce meth use and meth-associated sexual risk behavior. Ultimately, a pharmacologic treatment for meth use may not only serve to improve outcomes among those who are accessing current treatment services, but might also benefit those who are not willing or able to utilize such services. While studies show that MSM who enter substance use treatment decrease both their substance use and sexual risk behavior, current behavioral meth treatment programs report low rates of success in treating meth dependence among MSM. We believe the time has come to test the acceptability of pharmacologic interventions to reduce meth use among MSM, and to assess the feasibility of conducting such trials among sexually active, meth-dependent MSM, whose meth-associated sexual behavior use places them at extraordinarily high risk for transmitting or acquiring HIV. In this pilot study, we will provide meth-dependent MSM with placebo or daily bupropion XL (extended-release), a well-tolerated dopamine agonist that has potential to reduce meth use. The specific aims of this study are:

1. To assess the feasibility of enrolling and retaining meth-dependent MSM into a randomized, double-blind study of bupropion versus placebo with biologic (urine meth testing) and behavioral (sexual risk) measures.
2. To explore the tolerability of bupropion and placebo among meth-dependent MSM, as determined by the number of adverse clinical events in the bupropion and placebo arms.
3. To describe the acceptability of bupropion and placebo among meth-dependent MSM, by measuring (via electronic pill caps) medication adherence to bupropion and placebo.

This randomized, double-blind, placebo-controlled, two-arm pilot study will enroll 30 meth-dependent MSM assigned to receive 3 months of bupropion XL 300 mg daily or placebo. We will include both HIV- and HIV-INFECTED MSM, because meth use is common in both groups. We will enroll meth-dependent MSM because they are the most likely population to benefit from this potential treatment. Participants will be seen weekly for urine specimen collection and substance-use counseling. Clinical exams, medical history, specimen collection, and behavioral assessments will be performed at baseline and at the 1, 2, and 3 month visits. Interim visits will be scheduled whenever indicated by signs or symptoms. Our decision to maintain participants on 3 months of bupropion is based on the smoking literature, which demonstrated bupropion's efficacy in treating nicotine addiction within similar time periods; we anticipate that any future efficacy trial will maintain participants on bupropion for this duration.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative by rapid test or able to document HIV infection through healthcare provider's note or documentation of laboratory test;
* Reports anal sex with men in prior 3 months while using meth
* Diagnosed with meth dependence as determined by SCID
* Interested in stopping or reducing meth use
* Meth-positive urine on screening
* No known allergies to bupropion
* No current acute illnesses
* Able and willing to provide informed consent and to be followed over a 3-month period
* Baseline CBC and electrolytes within institutional limits.

Exclusion Criteria:

* History of seizure
* High risk for seizure, including: recent (last 24 months) head trauma, brain injury or surgery; using theophylline or systemic steroids; prior or current history of anorexia or bulimia; prior or current history of alcohol withdrawal symptoms
* Measured moderate or severe liver disease (LFTs > 3 times normal) or history of chronic liver disease
* Impaired renal function (creatinine clearance < 90 ml/min)
* Evidence of current major depression, as determined by SCID
* Taking anti-depressant medication within last 30 days
* Currently on any bupropion-containing regimen
* Currently using or unwilling not to use pseudoephedrine-containing products (causes false + urines for meth use) for trial duration
* Currently taking antiretroviral therapy (ART)
* CD4 count < 200 cells/mm3
* Any condition that, in the principal investigator's judgment, interferes with safe study participation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Colfax, M.D., Principal Investigator — Co-Director, HIV /AIDS Statistics, Epidemiology and Intervention Research Section
Locations (1):
- San Francisco Department of Public Health, HIV/AIDS Office, San Francisco, California, United States

REFERENCES:
- [Result] Das M, Santos D, Matheson T, Santos GM, Chu P, Vittinghoff E, Shoptaw S, Colfax GN. Feasibility and acceptability of a phase II randomized pharmacologic intervention for methamphetamine dependence in high-risk men who have sex with men. AIDS. 2010 Apr 24;24(7):991-1000. doi: 10.1097/qad.0b013e328336e98b. PMID 20397286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were actively recruited at the municipal STD and HIV clinics, and by street outreach. Recruitment flyers were posted at locations of active recruitment, in local newspapers and in print media and on social networking websites.
Pre-assignment Details: After informed consent, participants were screened in two screening visits, with lab and HIV testing, medical history and physical exam, and urine meth testing.
Groups:
- Bupropion: Bupropion XL 300mg daily
Period: Overall Study
Arm/Group | Bupropion | Placebo
Started | 20 | 10
Completed | 18 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Proportion of Persons Screened Who Are Eligible and Enrolled
Time Frame: At Enrollment
Measure: Number; unit: Eligible persons screened who enrolled
Arm/Group | Persons Screened
Number analyzed (Participants) | 54
Eligible persons screened who enrolled | 30

2. Primary Outcome: Feasibility: Proportion of Scheduled Study Visits Completed
Time Frame: 12 weeks
Measure: Number; unit: Scheduled study visits completed
Units Other Than Participants: Study visits after enrollment
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
Number analyzed (Study visits after enrollment) | 240 | 120
Scheduled study visits completed | 185 | 96

3. Primary Outcome: Feasibility: Proportion of Urine Samples Collected
Time Frame: 12 weeks
Measure: Number; unit: Urine samples collected
Units Other Than Participants: Study visits post enrollment
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
Number analyzed (Study visits post enrollment) | 240 | 120
Urine samples collected | 193 | 97

4. Primary Outcome: Feasibility: Participants Who Completed the Trial
Time Frame: 12 weeks
Measure: Number; unit: participants who completed the trial
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
participants who completed the trial | 18 | 9

5. Primary Outcome: Tolerability: Comparison of Adverse Events in the Bupropion and Placebo Arms.
Time Frame: throughout study
Measure: Number; unit: number of adverse events
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
number of adverse events | 40 | 11

6. Primary Outcome: Acceptability: Adherence to Daily Bupropion and Placebo, as Determined by MEMS (Medication Event Monitoring System) Caps Openings
Description: Proportion of days in which the MEMS cap device was opened during of the 12 weeks on study drug.
Time Frame: 12 weeks
Measure: Number; unit: percentage adherence by MEMS
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
percentage adherence by MEMS | 59 | 62
Statistical Analysis 1: Comparison: Bupropion vs Placebo; Test type: Superiority or Other; p = 0.98, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Acceptability: Adherence to Daily Bupropion and Placebo, as Determined by Self-report
Description: Proportional of reported days taking study drug during the 12 weeks of study.
Time Frame: 12 weeks
Measure: Number; unit: percentage of self-reported adherence
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
percentage of self-reported adherence | 85 | 75

8. Primary Outcome: Acceptability: Proportion of Participants Discontinuing Medication in Both Arms
Description: Proportion of participants who discontinued study medication for at least one week prior to study completion.
Time Frame: 12 weeks
Measure: Number; unit: percentage of discontinuations
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 20 | 10
percentage of discontinuations | 15 | 30

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 17/20 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=20) | Placebo (N=10)
Soft tissue infection (Infections and infestations) | 4 (5) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Stimulant toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Allergic reaction to antibiotics (Immune system disorders) | 1 (1) | 0 (0)
Decreased CD4 (Investigations) | 1 (1) | 0 (0)
Decreased libido (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Sexually transmitted infection (Infections and infestations) | 1 (1) | 1 (1)
HIV Seroconversion (Immune system disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Increased ALT (Hepatobiliary disorders) | 4 (5) | 2 (2)
Increased AST (Hepatobiliary disorders) | 3 (3) | 2 (2)
Increased creatinine (Renal and urinary disorders) | 3 (3) | 0 (0)
Sleep Disturbances (General disorders) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes